CLINICAL TRIAL: NCT05933967
Title: A Phase II, Prospective ,Multicenter Study Evaluating the Efficacy and Safety of Orelabrutinib Plus R-CHOP in Treatment-naïve Patients With Double Expression Diffuse Large B-cell Lymphoma
Brief Title: A Study of Orelabrutinib Plus R-CHOP in Treatment-naïve Patients With Double Expression Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Zengjun Li, Head of the Hematology Department, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDCHI-NHL-001
Record Dates: First submitted 2023-06-16; First posted 2023-07-06 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: The First Affiliated Hospital of Nanchang University

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- orelabrutinib+R-CHOP (Experimental)
  Interventions: Drug: Orelabrutinib+R-CHOP

INTERVENTIONS:
Drug: Orelabrutinib+R-CHOP — Orelabrutinib 150mg qd PO. Rituximab 375 mg/m2 IV on Day 0 of each 21-day cycle. The CHOP include cyclophosphamide, doxorubicin/Epirubicin/liposomal doxorubicin, vincristine/Vindesine, and prednison.

SUMMARY:
This is a multicenter prospective single arm phase II study, and the purpose of this study is to evaluate the safety and efficacy of orelabrutinib combined with R-CHOP in the treatment of treatment-naïve patients with double expression DLBCL.

DETAILED DESCRIPTION:
The patients will be treated with 6/8 cycles of orelabrutinib plus R-CHOP regimen（21 days per cycle). The primary objective was the complete response rate (CRR) at end of induction therapy

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Double Expression Diffuse Large B-cell Lymphoma

  * Age 18-70 years
  * ECOG performance status 0-2
  * Ann Arbor stage II-IV
  * 8.Subjects who in line with the testing standard of the clinical trial laboratory
  * Life expectancy ≥ 3months

Exclusion Criteria:

* • systemic lymphoma involved CNS.

  * Accompanied by uncontrolled cardiovascular and cerebrovascular diseases, coagulopathy, connective tissue diseases.
  * uncontrolled infections (including HBV, HCV, HIV/AIDS)
  * Subjects who prepared for transplantation
  * Pregnancy or active lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
complete response rate | up to 24 weeks

SECONDARY OUTCOMES:
ORR | up to 24 weeks
  ORR is defined as the proportion of patients with a best response of CR or PR
2 years progression-free survival | From date of receiving the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years]
  2 years progression-free survival was calculated from the date of therapy until death from lymphoma or 2-year follow-up without relapsing
2 years overall survival | From date of receiving the first dose until the date of death from any cause,assessed up to 2 years
  2 years overall survival was calculated from the date of therapy until death from lymphoma or 2-year follow-up alive
The occurrence of adverse events and serious adverse events | up to 30 months
  Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: zengjun Li, Study Chair — Shandong Cancer Hospital and Institute, Shandong First Medical University and Shandong Academy of Medical Sciences
Locations (2):
- China (2):
  - The First Ailliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shandong Cancer Hospital and Institute, Shandong First Medical University and Shandong Academy of Medical Sciences, Jinan, Shandong